CLINICAL TRIAL: NCT07328490
Title: A Phase I/II Study to Assess the Safety and Antitumor Activity of Bispecific T-cell Engager Tarlatamab and TROP2 Targeted Antibody Drug Conjugate Sacituzumab Govitecan in Previously Treated Extensive-Stage Small Cell Lung Cancer and Extrapulmonary Neuroendocrine Cancer
Brief Title: Bispecific T-Cell Engager Tarlatamab and TROP2 Targeted Antibody Drug Conjugate Sacituzumab Govitecan in Previously Treated Extensive-Stage Small Cell Lung Cancer and Extrapulmonary Neuroendocrine Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001942; 001942-C
Record Dates: First submitted 2026-01-08; First posted 2026-01-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-06

CONDITIONS: Extensive-Stage Small Cell Lung Cancer; Extrapulmonary Neuroendocrine Carcinoma; Small Cell Carcinoma
Keywords: Tarlatamab; Sacituzumab Govitecan; Bispecific T-cell Engager; Immunotherapy; Antibody Drug Conjugate; Targeted Therapy
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Small Cell | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/ Phase I (Experimental): Dose escalated Tarlatamab and Sacituzumab Govitecan
  Interventions: Drug: Tarlatamab; Drug: Sacituzumab Govitecan
- 2/ Phase II (Experimental): Maximum tolerated dose (MTD) Tarlatamab and Sacituzumab Govitecan
  Interventions: Drug: Tarlatamab; Drug: Sacituzumab Govitecan

INTERVENTIONS:
Drug: Tarlatamab — For both Phase I and Phase II, participants will receive a step dose of 1 mg of Tarlatamab (IV) followed by a full dose of 10 mg starting 7 days later (i.e., step dosing phase). Cycle 1 will begin following the Tarlatamab step-dosing (i.e., 14 days after the first dose and 7 days after the second dose of Tarlatamab alone) with participants receiving a combination of Tarlatamab (full dose) and Sacituzumab Govitecan (IV 7.5 or 10 mg/Kg) on day 1, SG alone on day 8 and Tarlatamab alone on day 15 of every cycle (4-week cycles) for up to 2 years or until disease progression/death, development of intolerable side effects.
Drug: Sacituzumab Govitecan — For both Phase I and Phase II, participants will receive a step dose of 1 mg of Tarlatamab (IV) followed by a full dose of 10 mg starting 7 days later (i.e., step dosing phase). Cycle 1 will begin following the Tarlatamab step-dosing (i.e., 14 days after the first dose and 7 days after the second dose of Tarlatamab alone) with participants receiving a combination of Tarlatamab (full dose) and Sacituzumab Govitecan (IV 7.5 or 10 mg/Kg) on day 1, SG alone on day 8 and Tarlatamab alone on day 15 of every cycle (4-week cycles) for up to 2 years or until disease progression/death, development of intolerable side effects.

SUMMARY:
Background:

Small-cell lung cancer (SCLC) is the most deadly form of lung cancer. It kills at least 250,000 worldwide each year. Extra-pulmonary neuroendocrine cancer (EP-NEC) is a similar type of cancer that develops anywhere other than the lungs. EP-NEC is also very aggressive. Better treatments are needed for these cancers.

Objective:

To test 2 drugs (tarlatamab combined with sacituzumab govitecan [SG]) in people with SCLC or EP-NEC.

Eligibility:

People aged 18 years and older with SCLC or EP-NEC that either did not respond to or returned after treatment.

Design:

Participants will be screened with a physical exam, blood tests, heart function testing, and imaging scans.

Both study drugs are given intravenously (through a needle in the arm). Participants will receive a small starter dose of tarlatamab (1 mg) 2 weeks before beginning regular treatment, followed by the full dose (10 mg) one week later. Treatment then follows a repeating 4-week cycle: tarlatamab (10 mg) on days 1 and 15, and sacituzumab govitecan (7.5 or 10 mg/kg) on days 1 and 8. Treatment continues for up to 2 years, unless the cancer worsens, the participant passes away, or side effects become too severe.

Participants will have regular check-ups including physical exams, blood tests, and imaging scans to monitor safety and treatment response. Blood and tumor samples will be collected for research purposes.

After stopping treatment, participants will return for a safety check at 30 days, then be contacted every 3 months to check on their health and survival. Those who stop treatment for reasons other than cancer progression will continue CT scans every 6 weeks until their disease progresses.

DETAILED DESCRIPTION:
Background:

* Small-cell lung cancer (SCLC) is the most fatal and metastatic form of lung cancer which kills at least 250,000 people globally each year including more than 30,000 in the United States. SCLC constitutes approximately 14% of all lung cancers.
* SCLC consists of tumor cells with neuroendocrine (NE) and non-neuroendocrine (non-NE) features. SCLC subtypes exhibit distinct therapeutic vulnerabilities. Immunogenic plasticity and Notch signaling of non-NE SCLC underlie their responses to immune checkpoint blockade. NE SCLC is characterized by replication stress, rendering them susceptible to deoxyribonucleic acid (DNA) repair-targeted agents.
* The inhibitory Notch delta-like ligand 3 (DLL3) is aberrantly expressed on the surface of up to 85% of SCLC, mostly NE cells and minimally expressed in normal tissues, making it a compelling therapeutic target for NE SCLC. Trophoblast cell-surface antigen 2 (TROP2) is a transmembrane glycoprotein aberrantly expressed in SCLC during its progression from NE to the non-NE cell state, making it a compelling therapeutic target of non-NE SCLC.
* Tarlatamab is a bispecific T cell engager (BiTE) molecule which binds DLL3 on cancer cells and cluster of differentiation 3 (CD3) on T cells leading to T cell-mediated tumor lysis. Sacituzumab govitecan (SG) is an antibody drug conjugate (ADC) carrying a topoisomerase 1 (TOP1) inhibitor SN-38 payload to cancer cells expressing TROP2.
* Extrapulmonary neuroendocrine cancers (EP-NEC) are rare and aggressive orphan cancers that share morphological and transcriptomic similarities and potentially therapeutic vulnerabilities with SCLC, with no standard treatments at relapse.
* In the current study, combination therapies targeting DLL3 and TROP2, using a combination of tarlatamab and sacituzumab govitecan will be evaluated as potential drivers of durable response in SCLC and EP-NEC.

Objectives:

Phase I:

-To determine the maximum tolerated dose (MTD) of bispecific T-cell engager tarlatamab and TROP2 targeted antibody drug conjugate sacituzumab govitecan in participants with previously treated relapsed SCLC or EP-NEC.

Phase II:

-To determine the clinical benefit in terms of objective response rates (ORR) in participants with previously treated relapsed SCLC or EP-NEC.

Eligibility:

->=18 years.

* Histologically or cytologically confirmed SCLC or EP-NEC that has progressed or recurred after at least one previous platinum-based regimen and immunotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less.

Design:

* This is a Phase I/II, open label clinical trial aimed at identifying the MTD of Sacituzumab govitecan in combination with tarlatamab and assessing the efficacy with respect to objective response rate in recurrent SCLC and EP-NEC.
* Participants will receive a step dose of 1mg tarlatamab 14 days prior to the first cycle followed by a full dose (10mg) starting a week later. Thereafter, tarlatamab will be administered on days 1 and 15 and sacituzumab govitecan (7.5 or 10 mg/Kg) will be administered on days 1 and 8 of every 4-week cycle. Treatment will be administered for up to 2 years or until disease progression/death or development of intolerable side effects (whichever occurs first).
* During treatment, participants will have clinical assessments, laboratory evaluations, and imaging studies for safety and response assessment. Blood and tumor samples will be collected for correlative studies at various timepoints.
* Participants will be followed for survival every 3 months following objective disease progression.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Must have histologically or cytologically confirmed SCLC or EP-NEC meeting the criteria below:

  * SCLC that has progressed or recurred after a combination of platinum-based regimen and immunotherapy. Participants may be eligible after treatment with chemo or immunotherapy alone if they were intolerant to one of the components. Participants with previously locally advanced SCLC who have completed definitive chemoradiation therapy, with or without surgical resection, and subsequently experienced disease progression or recurrence, are also eligible. OR
  * EP-NEC that has progressed or recurred after at least one prior chemotherapy.
* Must have measurable disease, per RECIST 1.1
* Age >=18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status <=2.
* Must have adequate organ and marrow function as defined below:

System/Laboratory Value

Hematological

* Hemoglobin/>=9 g/dL(a)
* Absolute neutrophil count/>= 1,500/mcL
* Platelets/>= 100,000/mcL

System/Laboratory Value

Hepatic

* Total bilirubin/within normal institutional limits
* AST (SGOT) and ALT (SGPT)/<= 2.5 X institutional ULN (<=5 X ULN for participants with liver metastases)

Renal

-Creatinine/ within normal institutional limits

OR

-Calculated (b) creatinine clearance (GFR can also be used in place of creatinine or CrCl)/>=60 mL/min for participant with creatinine levels above institutional normal

OR

Coagulation

* Prothrombin time (PT)/<=1.5 (SqrRoot) ULN unless participant is receiving anticoagulant therapy if PT or PTT is within therapeutic range of intended use of anticoagulants
* Partial thromboplastin time (PTT)/<=1.5 (SqrRoot) ULN unless participant is receiving anticoagulant therapy if PT or PTT is within therapeutic range of intended use of anticoagulants

ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase);

AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase);

GFR=glomerular filtration rate; ULN=upper limit of normal.

1. Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
2. Creatinine clearance (CrCl) should be calculated per institutional standard.

   * Individuals with neurologically stable brain metastases defined as asymptomatic metastasis, or treated metastasis having no evidence of progression or hemorrhage for at least 1 week after treatment (including brain radiotherapy) may be included. Individuals must be off any systemic corticosteroids for the treatment of brain metastases for at least 7 days prior to study drug initiation.
   * Individuals with human immunodeficiency virus (HIV) must be on effective antiretroviral therapy with undetectable viral load at screening.
   * Individuals with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load at screening.
   * Individuals with a history of hepatitis C virus (HCV) infection must have been treated and cured. Individuals with active HCV infection who are currently on treatment are eligible if they have an undetectable HCV viral load at screening.
   * Must agree to use an effective method of contraception (barrier, hormonal, intrauterine device [IUD], surgical sterilization, abstinence) during study treatment and for 3 months thereafter for males or 6 months for women of childbearing potential (WOCBP).
   * Willingness to discontinue nursing during study treatment and for 2 months after the last dose of study treatment.
   * Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Receiving any other investigational agents or concurrent systemic anti-cancer therapies. Any previous non-investigational treatment must be completed at least 2 weeks prior to study drug initiation.
* Requiring radiation therapy during study treatment. Radiation therapy may be allowed if needed for palliative/symptom control (e.g., bone metastasis) but must be completed at least 7 days before study drug initiation.
* Severe and unresolved active autoimmune inflammatory conditions.
* Pregnant women at screening.
* Requiring immunosuppressive agents with the exception of those required by protocol, treatment for adverse events, Central Nervous System (CNS) metastases corticosteroid replacement therapy.
* Require live and live-attenuated vaccines during study treatment with tarlatamab or within 4 weeks of first dose of tarlatamab. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed. However, intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines and are not allowed.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs or other agents used in study.
* Requiring treatment with inhibitors or inducers of UGT1A1 during the planned period of study treatment.
* QTc >= 470 msec or any conditions or factors that may increase the risk of QTc prolongation.
* Uncontrolled intercurrent illness, evaluated by medical history and physical exam which would potentially increase risk to the participant.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose (MTD) | Dose Limiting Toxicity (DLT) period (C1D1 through C1D28)
  The toxicities identified at each dose level will be reported, by dose level, type, and grade.
Phase II: Objective Response Rate (ORR) | Until disease progression
  In each of the two main cohorts, the fraction of participants who experience a partial response (PR) or complete response (CR) will be reported along with a 95% confidence interval.

SECONDARY OUTCOMES:
Safety | Study duration
  Toxicities identified at each dose level will be reported, by dose level, type, and grade.
Overall survival (OS) | Until death or study is stopped
  OS will be calculated from the on-study date until date of death, or 6 months after the last study participant goes off-treatment, whichever comes earlier.
Duration of response (DOR) and Progression free survival (PFS) | Until disease progression
  Duration of response will be calculated by the Kaplan-Meier method, starting at date response was identified until progression or the response is declared to have ended, if the participants have a PR or CR.PFS will be calculated from on-study date until date of progression or death without progression, using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Anish Thomas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review.
Supporting Information: Study Protocol
Time Frame: Data will be made available as soon as possible or at the time of associated publication, whichever comes first.
Access Criteria: Data from this study may be requested by contacting the PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001942-C.html